CLINICAL TRIAL: NCT06743295
Title: Evaluation of Artificial Intelligence Based Noise Reduction in Phonak Hearing Aid on Patients With Hearing Impairment and Cochlear Implants
Brief Title: AI Noise Reduction in Phonak Hearing Aids
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Aniket Saoji, Associate Professor of Otolaryngology, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-009408
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Hearing Loss
Keywords: hearing aid
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Hearing Aid only (Experimental): Patients with hearing impairment who do not have a Cochlear implant
  Interventions: Device: DEEPSONIC™ Deep Sound Optimized Neural Integrated Chip Artificial intelligence-based noise reduction
- Cochlear Implant with Hearing Aid (Experimental): Patients with hearing impairment who have a single-sided implant (using a hearing aid on the opposite ear)
  Interventions: Device: DEEPSONIC™ Deep Sound Optimized Neural Integrated Chip Artificial intelligence-based noise reduction

INTERVENTIONS:
Device: DEEPSONIC™ Deep Sound Optimized Neural Integrated Chip Artificial intelligence-based noise reduction — Participants with hearing loss will be fitted with the Phonak Audéo Sphere™ Infinio (PAI) hearing aid with artificial intelligence (AI)-based noise reduction, which incorporates deep neural networks (DNN) technology to reduce background noise.
  Speech stimuli, presented at a comfortable level of approximately 60 dB SPL (like normal conversation), will be delivered via a loudspeaker positioned directly in front of the participant.
  They will be tested in 3 listening environments: quiet, moderate noise, high noise.
  Speech perception scores will be measured as a function of each hearing aid program setting: quiet setting, moderate noise, and advanced AI-based reduction for high noise.

SUMMARY:
The purpose of this study is to determine if artificial intelligence- based noise reduction can offer objective improvement in hearing and speech perception for hearing impaired patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hearing impairment not using hearing aids
* Individuals with hearing impairment currently using hearing aids
* Cochlear implant patients with a single-sided implant (using a hearing aid in the opposite ear)

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-04-24 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Single-word Testing | Baseline
  Participants will listen to a list of 50 words and repeat each word aloud. Results are reported as a percentage of correctly repeated words out of 50.
Sentence Testing | Baseline
  Participants will listen to a list of 20 sentences and repeat each sentence aloud. Results are reported as a percentage of correctly repeated sentences out of 20.

CONTACTS AND LOCATIONS:
Overall Officials: Aniket Saoji, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials